CLINICAL TRIAL: NCT02509091
Title: Clinical Efficacy and Safety of Therapy of Bronchoalveolar Lavage and Local Amikacin Injection in Patients With Acute Exacerbation of Bronchiectasis:An Open-label Randomized Parallel Controlled Study
Brief Title: Therapy of Bronchoalveolar Lavage and Local Amikacin Injection in Patients With Acute Exacerbation of Bronchiectasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Director, Head of respiratory medicine, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150616
Record Dates: First submitted 2015-07-22; First posted 2015-07-27 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The experimental group (Experimental): fundamental treatment combining with the therapy of bronchoalveolar lavage and local Amikacin injection.(fundamental treatment including anti-infection,eliminating phlegm,oxygen therapy etc.)
  Interventions: Drug: Bronchoalveolar Lavage and Local Amikacin Injection
- The controlled group (No Intervention): fundamental treatment(including anti-infection,eliminating phlegm,oxygen therapy etc.)

INTERVENTIONS:
Drug: Bronchoalveolar Lavage and Local Amikacin Injection — injecting 0.4g of AK in 100 ml to 250 ml, not exceeding 300 ml. And generally, repeat it for 3 to 5 times.
  Other Names: Amikin;AMK
  Arms: The experimental group

SUMMARY:
The therapy of bronchoalveolar lavage and local amikacin injection as one of the treatment of bronchiectasis developed in recent years.this study is aim to evaluate the Clinical Efficacy and Safety of Therapy of Bronchoalveolar Lavage and Local Amikacin Injection in Patients with Acute Exacerbation of Bronchiectasis.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the efficacy and safety of The therapy of bronchoalveolar lavage and local amikacin injection through the observation of a large sample of clinical cases. During the observation, study visits will occur at the end of 30days, 60days, 90days.all the participants will be required to check the various efficacy and safety indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years and ≤80 years;
2. Patients with non-cystic fibrosis bronchiectasis diagnosed by high-resolution CT;
3. Are sensitive to amikacin;
4. Acute exacerbation of bronchiectasis;
5. Capable of the completion of bronchoscopy, alveolar lavage, pulmonary function testing etc;
6. Willing to join in and sign the informed consent form.

Exclusion Criteria:

1. Active bleeding without control；
2. Receiving nasal or facial surgery recently；
3. With severe cardio-pulmonary dysfunction, such as left heart failure, unstable arrhythmia, etc.
4. With other respiratory diseases: such as active pulmonary tuberculosis, non-tuberculosis mycobacteria (NTM) pulmonary disease, pulmonary aspergillosis, etc.
5. Be allergic to amikacin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Improvement of Sputum volume and properties | 90 days
  Phlegm improvement will be measured by the reduction of the sputum volume and change of sputum properties in the first day,in admission,the first day before,in and after doing bronchoscopy ,the day in discharge and in 30 days/60 days/90 days

SECONDARY OUTCOMES:
changes in lung function (including Forced expiratory volume in one second (FEV1) ,forced vital capacity(FVC) and forced vital capacity rate of one second(FEV1/FVC)) | 90 days
  Lung function will be measured as improved/stabilized/exacerbated from baseline to 30 days/60 days/90 days
Dyspnea score according by Modified Medical Research Center(MMRC) | 90 days
  to measure rating dyspnea according by Medi Medical Research Center(MMRC) from baseline to 30 days/60 days/90 days
Cough score according by Leicester Cough Questionnaire(LCQ) | 90 days
  to measure rating cough according by Leicester Cough Questionnaire(LCQ) from baseline to 30 days/60 days/90 days
Life quality: assessed by St. George respiratory questionnaire (SGRQ) | 90 days
  Life quality will be assessed as improved if SGRQ single or total score increased >4% when completing the trial; stabilized if SGRQ single or total score changes within the range of 4% when completing the trial; exacerbated if SGRQ single or total score decreased >4% when completing the trial from baseline to 30 days/60 days/90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Fu Xu, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided